CLINICAL TRIAL: NCT04837443
Title: The Effect of the Rubber Hand Illusion on Sensory Thresholds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zafer Günendi, professor doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 217
Record Dates: First submitted 2021-03-18; First posted 2021-04-08 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: sensory threshold; rubber hand illusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous working group (Experimental)
  Interventions: Behavioral: Rubber hand illusion
- Asynchronous working group (Sham Comparator)
  Interventions: Behavioral: Rubber hand illusion

INTERVENTIONS:
Behavioral: Rubber hand illusion — Tactile sensory threshold from quantitative sensory tests, two point discrimination from cortical senses, pressure pain threshold measured by algometer will be examined during and after the rubber hand burning, which causes changes in body perception.

SUMMARY:
The rubber hand illusion (RHI) causes a change in body perception and awareness as a result of the integration of simultaneously perceived visual and tactile stimulation. In the rubber hand illusion (RHI), which was first described in 1998, a realistic hand model is perceived as a part of the body and body awareness is impaired. In the RHI, the participant's real hand is positioned behind a screen so that it is out of sight; The rubber model hand is placed in the field of vision and in the appropriate position with the real hand. Brush is applied simultaneously to the same parts of the real and rubber hands. He/she perceives the rubber hand as his own and the brush starts to feel as if it is being rubbed into his own hand. This method, which causes the illusion of body belonging, has been defined as the rubber hand illusion. During the rubber hand illusion, increased activity was observed in the ventral premotor cortex, infraparietal cortex and cerebellum in functional MRI. It is suggested that this phenomenon occurs with the integration of interrelated visual, tactile and proprioceptive senses reaching the premotor cortex.

Quantitative sensory tests are standardized subjective clinical sensitivity tests that require the collaboration of the person to be examined. In the tests, calibrated stimuli are applied to capture perception and pain thresholds, thus providing information about sensory thresholds.

The impairment of body perception caused by RHI contributes to the multi-faceted understanding of sensory perception, higher-level cognitive processes, brain mapping and functions. In the studies; It has been suggested that the conflict between visual and proprioceptive sensory information created during the rubber hand illusion is resolved by the attenuation of somatosensory input at the cortical level.

As far as we know, tactile sensory threshold from quantitative sensory tests, two-point discrimination from cortical senses, pressure pain threshold measured by the algometer, and vibration threshold variation during and after rubber hand burning, which causes changes in body perception, have not been studied before. In this study, the relationship between the RHI phenomenon and sensory thresholds will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18-65 years old age

Exclusion Criteria:

* Neuropathy
* Presence of any known neurological or psychiatric disease
* Inability to cooperate with the tests to be performed
* Amputation and nerve damage in the upper extremities
* Upper extremities dysfunction due to nerve damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
tactile sensation threshold | one hour
  Semmes-Weinstein monofilaments (SWM) are widely used for reproducible testing and measurement of tactile sensory threshold. The sizes of Semmes-Weinstein monofilaments increase on a logarithmic scale. It is made with nylon (line) monofilaments of approximately the same length. To apply, monofilaments are kept perpendicular to the skin and brought into contact. When the pressure is increased and the end point of the filament reaches the forcing threshold, the filament bends. Even if pressure is continued after the filaments are bent, there is no increase in the pressure felt on the skin. For this reason, when the monofilaments are inclined, since no more pressure can be applied with that filament, it is questioned whether the patient is felt or not. Three applications should be made to the patient with the same filament.
two point discrimination | one hour
  Two point discrimination (TPD) is the ability to distinguish between two points that are brought into contact with the skin at the same time and with the same pressure, that they are actually two separate points, not one. It was described by Ernest Heinrich Weber (1846). Blunt tip static and mobile TPD is usually tested using Disk-Criminator. Two points are brought into contact with the skin with a compass-like instrument or a compass. It can randomly switch between touching and touching a point or two points in the area being tested. The person being tested is asked to say how many points he felt. The smallest distance resulting in the perception of two different stimuli is recorded as the patient's two point discrimination threshold.
pressure pain threshold | one hour
  Pain pressure threshold is defined as the minimum pressure value that creates a perception of pain. The test determines the amount of pressure in a particular area as soon as an ever-increasing painless pressure stimulus turns into a painful feeling of pressure. The pressure algometer (dolorimeter) used for this test is a device used to evaluate sensitivity to pain. The mechanical method using the pressure sensor provides ease of use, is harmless to the patient, and has acceptable reliability and repeatability. Light pressure is applied to the body area to be tested with the algometer. The intensity of the pressure is increased gradually. The participant is asked to say the moment he feels the sensation of pain instead of pressure during the algometric measurement. The amount of pressure that causes pain is recorded as the pressure pain threshold (PPT) in kg / cm2. It has been shown that 3 measurements are required to maximize measurement properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine Department of PMR, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study is planned as a specialist thesis, the details of the study can be shared by the faculty administration.

REFERENCES:
- [Background] Tsakiris M, Prabhu G, Haggard P. Having a body versus moving your body: How agency structures body-ownership. Conscious Cogn. 2006 Jun;15(2):423-32. doi: 10.1016/j.concog.2005.09.004. Epub 2005 Dec 15. PMID 16343947
- [Background] Botvinick M, Cohen J. Rubber hands 'feel' touch that eyes see. Nature. 1998 Feb 19;391(6669):756. doi: 10.1038/35784. No abstract available. PMID 9486643
- [Background] Ramakonar H, Franz EA, Lind CR. The rubber hand illusion and its application to clinical neuroscience. J Clin Neurosci. 2011 Dec;18(12):1596-601. doi: 10.1016/j.jocn.2011.05.008. Epub 2011 Oct 13. PMID 22000838
- [Background] Mohan R, Jensen KB, Petkova VI, Dey A, Barnsley N, Ingvar M, McAuley JH, Moseley GL, Ehrsson HH. No pain relief with the rubber hand illusion. PLoS One. 2012;7(12):e52400. doi: 10.1371/journal.pone.0052400. Epub 2012 Dec 20. PMID 23285026
- [Background] Fang W, Zhang R, Zhao Y, Wang L, Zhou YD. Attenuation of Pain Perception Induced by the Rubber Hand Illusion. Front Neurosci. 2019 Mar 22;13:261. doi: 10.3389/fnins.2019.00261. eCollection 2019. PMID 30967758
- [Background] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Background] Won SY, Kim HK, Kim ME, Kim KS. Two-point discrimination values vary depending on test site, sex and test modality in the orofacial region: a preliminary study. J Appl Oral Sci. 2017 Jul-Aug;25(4):427-435. doi: 10.1590/1678-7757-2016-0462. PMID 28877282
- [Background] Haloua MH, Sierevelt I, Theuvenet WJ. Semmes-weinstein monofilaments: influence of temperature, humidity, and age. J Hand Surg Am. 2011 Jul;36(7):1191-6. doi: 10.1016/j.jhsa.2011.04.009. PMID 21712138